CLINICAL TRIAL: NCT05976204
Title: Prognostic Value of Neutrophil-Lymphocyte Ratio (NLR), Absolute Lymphocyte Count (ALC), and Thrombocyte-Lymphocyte Ratio (TLR) in Predicting the Outcomes of Tetralogy of Fallot Primary Repair
Brief Title: Prognostic Value of NLR, TLR, and ALC in Predicting ToF Primary Repair Outcome
Status: Completed | Type: Observational
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Sisca Natalia Siagian, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Other Study IDs: LB.02.01/VII/2023/NLR
Record Dates: First submitted 2023-07-14; First posted 2023-08-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Disease; Tetralogy of Fallot; Neutrophil-lymphocyte Ratio; Absolute Lymphocyte Count; Thrombocyte-lymphocyte Ratio; Outcome; TOF
Keywords: Congenital Heart Disease; Tetralogy of Fallot; Neutrophil-lymphocyte ratio; Absolute lymphocyte count; Thrombocyte-lymphocyte ratio; Outcome
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ToF primary repair: Patients who underwent ToF primary repair from January 2020 until December 2022
  Interventions: Procedure: ToF primary repair

INTERVENTIONS:
Procedure: ToF primary repair — ToF primary repair for patients with ToF

SUMMARY:
Tetralogy of Fallot (ToF) were cyanotic congenital heart disease with chronic hypoxia which increases the risk of exacerbated inflammatory response in ToF primary repair. Various studies have recently shown inflammatory biomarkers to predict morbidity and mortality in hypoxemic patients, but they are not readily available and expensive.This study aims to compare the prognostic value of neutrophil-lymphocyte ratio (NLR), absolute lymphocyte count (ALC), and thrombocyte-lymphocyte ratio (TLR) in predicting ToF primary repair outcomes. This was a retrospective observational study on ToF primary repair in National Cardiovascular Center Harapan Kita between Januari 2020 until December 2022. Preoperative NLR, ALC, and TLR were derived from blood test obtained <14 days before surgery. The primary endpoints were redo surgery, 30-day mortality, and complications. The secondary endpoints were hospital length of stay (HLOS) and postoperative LOS.

DETAILED DESCRIPTION:
This was a retrospective observational study on tetralogy of Fallot (ToF) primary repair in National Cardiovascular Center Harapan Kita between Januari 2020 until December 2022. The preoperative demographic data included were patients' gender, age, weight, oxygen saturation, and associated diagnosis other than ToF. The preoperative data of complete blood count and differential count must be tested from the most recent peripheral blood samples taken no later than 14 days before the surgery. The data obtained were the number of days of the most recent blood test including the leukocyte count, percentage neutrophil, percentage and absolute lymphocyte count, thrombocyte count, as well as the derived variables such as neutrophil lymphocyte ratio (NLR) ratio and thrombocyte lymphocyte ratio (TLR). The intraoperative data included were the use of cardiopulmonary bypass (CPB), CPB time, aortic cross-clamp (AOX) time, and the total duration of surgery. Patients were evaluated and followed-up for any complications and postoperative mortality during the same hospital stay until discharge. Patients were then followed up for any cause of mortality within 30 days postoperative.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ToF and any other associated cardiac anomalies, who underwent ToF primary repair and had a complete blood cell count with differential count available preoperatively

Exclusion Criteria:

* Surgery other than ToF primary repair
* Association with other procedures (except patent ductus arteriosus/PDA ligation, patent foramen ovale/PFO or atrial septal defect/ASD closure, or pulmonary arteries enlargement)
* Preoperative hemodynamic instability
* Suspected or confirmed infection with prior antibiotic administration during the same hospital admission
* Absence of complete blood count with differential count

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients who underwent ToF primary repair in National Cardiovascular Center Harapan Kita between Januari 2020 until December 2022
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients Requiring Redo surgery | From the initial primary ToF until the discharge of the patients or until 2 weeks after the operation, whichever came first
  Redo surgery was defined as additional or corrective surgery after the initial primary ToF repair within the same hospital admission.
Mortality | Until 30 days postoperative
  Mortality intraoperative or postoperative
Complications (categorized as mild, moderate, severe) | From the initial primary ToF until the discharge of the patients or until 2 weeks after the operation, whichever came first
  Complication was defined as any adverse events that arised during the operation or postoperative until the discharge of the patient.

SECONDARY OUTCOMES:
Hospital Length of Stay | From the initial primary ToF until the discharge of the patients or until 12 weeks after the operation, whichever came first
  Hospital length of stay (HLOS) was defined as the duration of stay in the hospital from the initial admission to discharge.
Postoperative Length of Stay | From the initial primary ToF until the discharge of the patients or until 12 weeks after the operation, whichever came first
  Longer postoperative LOS was defined as hospitalization of more than 5 days from the period of surgery until postoperative discharge (based on our center).

CONTACTS AND LOCATIONS:
Overall Officials: Sisca N Siagian, MD, Principal Investigator — National CCHK
Locations (1):
- National Cardiovascular Center Harapan Kita Jakarta Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
At the moment, the investigators have no plan to share the whole participant data. However, if it is needed, the investigators will

REFERENCES:
- [Derived] Siagian SN, Christianto C. Prognostic value of neutrophil-lymphocyte ratio, absolute lymphocyte count, and thrombocyte-lymphocyte ratio in predicting the outcomes of tetralogy of fallot primary repair. Front Cardiovasc Med. 2025 Jun 5;12:1489242. doi: 10.3389/fcvm.2025.1489242. eCollection 2025. PMID 40538915